CLINICAL TRIAL: NCT03844516
Title: Work Intolerance in Left Ventricular Assist Device Recipients: Impact of Pacing
Brief Title: Pacing in Left Ventricular Assist Device Recipients
Acronym: Pace-VAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Finn Gustafsson (Other)
Responsible Party: Sponsor-Investigator, Finn Gustafsson, Professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: H-17029488
Record Dates: First submitted 2019-02-15; First posted 2019-02-18 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Heart Rate; Chronotropic Incompetence; Pacing
Keywords: Chronotropic incompetence; pacing; heart rate; exercise; peak oxygen uptake
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Patients and staff performing the peak oxygen uptake test (pVO2) will be blinded to device regulation. Blinding will be ensured by recruiting a secondary doctor or other staff to regulate pace-settings in relation to the paced pVO2 test while performing sham regulations (or just read pace-settings) in relation to the non-paced pVO2 test.
  Thus, both patients and investigator are blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peak oxygen uptake test with pacing (Other): Peak oxygen uptake test with pacing
  Interventions: Other: Peak oxygen uptake test with pacing
- Peak oxygen uptake test without pacing (Sham Comparator): Peak VO2 test without pacing
  Interventions: Other: Peak oxygen uptake test without pacing

INTERVENTIONS:
Other: Peak oxygen uptake test with pacing — Peak oxygen uptake test with paced heart rate
  Other Names: Regulation of pace-device
  Arms: Peak oxygen uptake test with pacing
Other: Peak oxygen uptake test without pacing — Peak oxygen uptake test without paced heart rate
  Other Names: Sham pacing
  Arms: Peak oxygen uptake test without pacing

SUMMARY:
Implantation with left ventricular assist device (LVAD) in patients with end-stage heart failure (HF) leads to improvements in survival and quality of life, however, work capacity remains disappointingly low, at half of the expected value. Complex central and peripheral hallmarks of heart failure attribute to the continued work intolerance, to which heart rate may be a contributing factor.

The purpose of this study is to clarify the impact of heart rate (by means of pacing) on work capacity (measured as peak oxygen uptake) in LVAD recipients.

DETAILED DESCRIPTION:
While implantation with left ventricular assist devices (LVADs) in patients with end-stage heart failure (HF) improve survival and quality of life, work capacity remains at a disappointing 50% of the expected value.

Due to the worldwide (increasing) shortage of donor hearts, LVADs are increasingly used as destination therapy which makes it crucial for physicians to persistently identify opportunities to improve management, lower the adverse events and maximize the benefits of this treatment option.

In recent years it was found that upregulation of device pump speed improves the maximal work capacity of LVAD recipients with no side effects. More recently it was found that the patients' heart rate reserve also was of importance in this regard, however, the latter was shown in a retrospective study and needs to be confirmed in a prospective randomized double-blinded intervention study. As a large portion of LVAD recipients are already implanted with a pacing device (and suffer from chronotropic incompetence) such a study is possible to conduct by controlling their heart rate during exercise by pacing (ie randomized crossover design).

ELIGIBILITY:
Inclusion Criteria:

* Implanted with a left ventricular assist device
* Implanted with a pace-device ensuring the possibility of pacing
* Age > 18

Exclusion Criteria:

* Not able to undergo a peak oxygen uptake test
* No consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-04-23 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Peak oxygen uptake (pVO2) | 1 Day

SECONDARY OUTCOMES:
Heart rate | 1 Day

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, DK, Denmark